CLINICAL TRIAL: NCT01907659
Title: Viral Testing and Biomarkers to Reduce Antibiotic Use for Respiratory Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Rochester General Hospital (Other)
Responsible Party: Principal Investigator, Ann Falsey, Professor of Medicine, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABX RED-001; RGH KIDD-001 (Other: Rochester General Hospital KIDD Fund)
Record Dates: First submitted 2013-06-27; First posted 2013-07-25 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Respiratory Infections
Keywords: Respiratory; Viruses; Bacterial; Antibiotics; Procalcitonin
MeSH Terms: conditions — Respiratory Tract Infections; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of care (No Intervention): Standard of care for respiratory infections
- Release of test results (Experimental): Health care providers will receive viral PCR and PCT test results along with an algorithm recommending antibiotic treatment based on PCT level.
  Interventions: Other: Release of test results

INTERVENTIONS:
Other: Release of test results — Subjects will be randomized to have viral testing and serum PCT results released or no additional testing performed other than that ordered as standard of care
  Other Names: Viral PCR; Serum Procalcitonin
  Arms: Release of test results

SUMMARY:
This trial is a pilot study to determine the feasibility of a randomized clinical trial comparing a treatment algorithm consisting of a limited number of clinical parameters, rapid molecular viral diagnostics, and serum procalcitonin testing to standard of care for directing antibiotic use in patients with non-pneumonic lower respiratory tract infection. The reduction in antibiotic use in those subjects randomized to the treatment algorithm compared to those randomized to standard care will be determined.

DETAILED DESCRIPTION:
This is trial is a pilot study to determine the feasibility of a randomized clinical trial comparing a treatment algorithm consisting of a limited number of clinical parameters, rapid molecular viral diagnostics, and serum procalcitonin testing to standard of care for directing antibiotic use in patients with non-pneumonic lower respiratory tract infection. The reduction in antibiotic use in those subjects randomized to the treatment algorithm compared to those randomized to standard care will be determined. In addition, the added benefit of viral diagnosis to that of serum procalcitonin alone in reducing antibiotics will be determined. Lastly, antibiotic related complications and clinical outcomes to determine the safety of this approach at 30 days and 3 months in the standard care and intervention group will be evaluated. Analysis of the composite adverse event outcome (death, intensive care unit transfer, disease specific complications and recurrent respiratory tract infection requiring hospitalization) will serve as the principle safety analysis for the study. In addition, each adverse outcome will be examined individually as well as lesser adverse outcomes including antibiotic prescriptions, time to return to baseline health, patient reported outcomes and functional status at 30 days and 3 months. Physicians will be queried to determine factors which drive antibiotic prescriptions and potential barriers to implementing antibiotic reduction algorithms. These data will be used to design a phase III clinical trial with the intent to demonstrate that physicians in the US will respond appropriately to this information and that antibiotic use can be significantly and safely curtailed.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with symptoms of a respiratory infection
* Age > 21 years
* Systolic Blood Pressure > 90mm Hg
* Patient or health care designee can provide written informed consent

Exclusion Criteria:

* Intensive Care Requirement
* Antibiotics received prior to admission
* More than 24 hours of antibiotics received prior to enrollment
* Active chemotherapy or pulmonary radiation therapy
* Immunosuppressive conditions
* Conditions know to increase PCT values
* Definite infiltrate on CXR •% of band forms in peripheral blood > 15

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Antibiotic days | Total antibiotic days within 30 days after randomization
  The primary patient-level outcome is the number of days on antibiotics after randomization. The primary null hypothesis is that the distribution of the number of days on antibiotics is identical for the standard-of-care versus intervention arm, where the latter includes those patients for whom the PCT-intervention recommendation was overruled by the care team.

SECONDARY OUTCOMES:
Composite adverse events at 30 days and 3 months | 30 days and 3 months
  The secondary analyses will compare the following outcome variables between the intervention and the standard care group. Outcome variables will include total antibiotic related complications, length of hospitalization, a composite of 30 day and 3 month adverse events (death, ICU transfer, disease specific complications [development of pneumonia, lung abscess, empyema or ARDS] and recurrent LRTI requiring hospitalization).

OTHER OUTCOMES:
Physician attitudes regarding antibiotic prescription | 24 hours after release of intervention test results
  Physicians will be queried 24 hours after release of intervention results of viral testing and PCT values to understand factors associated with continuing or stopping antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: Ann R Falsey, MD, Principal Investigator — University of Rochester
Locations (1):
- Rochester General Hospital, Rochester, New York, United States

REFERENCES:
- [Derived] Branche AR, Walsh EE, Vargas R, Hulbert B, Formica MA, Baran A, Peterson DR, Falsey AR. Serum Procalcitonin Measurement and Viral Testing to Guide Antibiotic Use for Respiratory Infections in Hospitalized Adults: A Randomized Controlled Trial. J Infect Dis. 2015 Dec 1;212(11):1692-700. doi: 10.1093/infdis/jiv252. Epub 2015 Apr 24. PMID 25910632